CLINICAL TRIAL: NCT00478855
Title: Association of Antibiotic Utilization Measures and Control of ESBLs Producing Bacteria
Brief Title: Tazocin Intervention Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0910X-102105
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Piperacillin, Tazobactam Drug Combination; Piperacillin

INTERVENTIONS:
Drug: Tazocin (Piperacillin/Tazobactem)

SUMMARY:
1. To determine the value of using piperacillin/tazobactam in reducing the cases of extended spectrum beta lactamases (ESBL) producing E. coli or K. pneumoniae colonization and infection.
2. To determine the acquisition rate of ESBL producing E. coli or K. pneumoniae, both pre-and post-intervention in the selected medical centers.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted or transferred to the ICU/pulmonary/Infection units
* Patients of either sex, 18 years of age or older Patients who stay in units less than 48 hours will not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2006-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The acquisition rate of ESBL producing E. coli or K. pneumoniae at the end of phase I (pre-intervention) and phase II (last 3 months; post-intervention)

SECONDARY OUTCOMES:
The infection rate due to ESBL producing E. coli or K. pneumoniae at the end of phase I (pre-intervention) and phase II (last 3 months; post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Beijing, China